CLINICAL TRIAL: NCT03442673
Title: A Randomized Phase II Trial Comparing Stem Cell Mobilization With Chemotherapy and Cytokine (G-CSF) Versus Cytokine (G-CSF) Alone in Myeloma Patients (MOCCCA-trial).
Brief Title: Chemotherapy and G-CSF for Mobilization
Acronym: MOCCCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOCCCA-Trial
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Vinorelbine; Gemcitabine; G-CSF; ASCT
MeSH Terms: conditions — Multiple Myeloma | interventions — Vinorelbine; Gemcitabine; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CG (Chemotherapy/G-CSF) - Regime (Active Comparator): Vinorelbine 35 mg/m2 at day 1 as an i.v. infusion over 10 minutes or gemcitabine 1250 mg/m2 as a 30 minutes infusion at day 1. G-CSF will be started at day 4 at 10mcg/kg b.w. split in two daily doses, until the end of the stem cell collection procedure, with the first collection attempt on day 8.
  Interventions: Drug: Vinorelbine; Drug: Gemcitabine; Drug: G-CSF
- G (G-CSF) - Regime (Experimental): G-CSF at 10mcg/kg b.w. split in two daily doses starting from day 1 until the end of the stem cell collection procedure, with the first collection attempt on day 5.
  Interventions: Drug: G-CSF

INTERVENTIONS:
Drug: Vinorelbine — Stimulation with vinorelbine together with G-CSF for mobilization of autologous stem cells
  Arms: CG (Chemotherapy/G-CSF) - Regime
Drug: Gemcitabine — Stimulation with gemcitabine together with G-CSF for mobilization of autologous stem cells
  Arms: CG (Chemotherapy/G-CSF) - Regime
Drug: G-CSF — Cytokine stimulation with G-CSF for mobilization of autologous stem cells

SUMMARY:
This study aims to demonstrate that the mobilization with cytokine stimulation with G-CSF alone is non-inferior as compared to the standard mobilization with chemotherapy and G-CSF while associated with fewer side effects in myeloma patients.

DETAILED DESCRIPTION:
Background and Rationale High-dose chemotherapy (HDCT) with melphalan and autologous stem cell transplantation (ASCT) remains an integral component of the myeloma treatment algorithm for patients considered eligible for the procedure, nowadays performed in myeloma patients up to the age of 75 years. Until the advent of the novel agents, the initial therapy regimens commonly used were vincristine, doxorubicin, and dexamethasone (VAD) or single-agent dexamethasone, both of which shared the advantage of having little impact on stem cell mobilization and collection. Previous studies had shown that alkylating agents can potentially affect the stem cell pool and thus interfere with the ability to collect adequate numbers of stem cells. However, VAD is no longer uses nowadays, whereas current lenalidomide-containing combinations significantly affect stem cell collection. .In Switzerland, the combination of non-myeloablative chemotherapy with vinorelbine or gemcitabine and G-CSF is the current standard procedure. With the predominant use of bortezomib during induction treatment more patients have pre-existing neurotoxicity. Vinorelbine can aggravate this problem. Recently data have shown that a mobilization with gemcitabine together with G-CSF is safe and effective in myeloma patients. Whether chemotherapy is mandatory at all to achieve the same reliable and cost-effective mobilization is currently unknown. The investigators therefore consider that a direct comparison between vinorelbine/gemcitabine and G-CSF versus G-CSF alone is justified.

Objective:

The primary objective is to show non-inferiority of cytokine stimulation with G-CSF compared to chemotherapy stimulation with vinorelbine (or gemcitabine) together with G-CSF for the mobilization of autologous stem cells in myeloma patients in first remission.

Study Duration:

The anticipated total study duration is 42 months.

ELIGIBILITY:
Inclusion Criteria:

* Myeloma or amyloidosis patients after standard first-line induction treatment. (Additional induction regimens in refractory myeloma patients are allowed)
* Patients must be considered being clinically fit for subsequent consolidation with high-dose melphalan-based chemotherapy with autologous stem cell support.
* Patients must be aged ≥18 years.
* Female patients of child-bearing potential must have a negative pregnancy test (urine or serum) within 14 days prior to study treatment mobilisation, and they must implement adequate measures (hormonal treatment p.o. or i.m., intra uterine surgical devices, or latex condoms) to avoid pregnancy during study treatment and for additional 12 months.
* Patients must have given voluntary written informed consent

Exclusion Criteria:

* Patients with concurrent other malignant disease can be included, but previous treatment for other malignancies must have been terminated at least 2 months before registration. Endocrine treatment (such as for breast cancer) is allowed.
* Pregnancy or lactating female patients.
* The use of any anti-cancer investigational agents within 14 days prior to the expected start of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Number of patients achieving a sufficient number of stem cells | 8 days
  Number of patients achieving a sufficient number (at least 5.0 Mio/kg) of stem cells at the planned day in a single day procedure without the use of the rescue compound plerixafor

SECONDARY OUTCOMES:
Adverse events | 30 days after ASCT
  Number of patients experiencing toxicities/adverse events assessed according to the CTCAE 5.0 during the study period
Quality of life | 8 days
  Assessment of quality of life before and after mobilization. The EORTC Q30 questionnaire will be given to patients at screening and after mobilization
Pain | 8 days
  Assessment of pain associated with the mobilization procedure. Pain is measured with visual analogue scale before and after mobilization
Use of plerixafor | 8 days
  Number of patients requiring plerixafor for mobilization
Hematologic engraftment after ASCT | 30 days
  First day (after ASCT) of neutrophils rising again above 0.5 G/l, and of platelets rising again above 20 G/L in the absence of platelet transfusions in the previous 3 days.
Cellular composition of the peripheral blood and the grafts | 30 days
  Standard multiparameter flowcytometric assessment will determine CD4, CD8, sCD3, CD56 and CD19 cellular subsets.
Flowcytometric MRD levels in the peripheral blood and the grafts | 30 days
  Assessed by standard multiparameter flowcytometry.
Overall survival | 60 months
  Time from ASCT until death of any cause or date of last follow-up.
Progression free survival | 60 months
  Time from ASCT until first recurrence of myeloma or date of last follow-up whatever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Jeker, MD, Study Chair — Department for Medical Oncology University Hospital/Inselspital 3010 Bern Switzerland
Locations (1):
- Department for Medical Oncology University Hospital/Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Jeker B, Thalmann L, Bacher U, Nilius H, Rhyner G, Sokler M, Soltermann S, Winkler A, Vorburger C, Daskalakis M, Hoffmann M, Pabst T. Comparing stem cell mobilization with chemotherapy and cytokine (G-CSF) versus cytokine alone in myeloma patients (MOCCCA): a randomized phase II, open-label, non-inferiority trial. Bone Marrow Transplant. 2025 Mar;60(3):270-276. doi: 10.1038/s41409-024-02468-z. Epub 2024 Nov 15. PMID 39548306